CLINICAL TRIAL: NCT01858402
Title: The Efficacy of Intravenous Paracetamol Versus Dipyrone for Postoperative Analgesia After Day-case Lower Abdominal Surgery in Children With Spinal Anesthesia: a Prospective Randomized Double-blind Study
Brief Title: Paracetamol Versus Dipyrone After Pediatric Lower Abdominal Surgery in Children With Spinal Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Esra Caliskan, Associated Professor, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KA 09/06
Record Dates: First submitted 2013-05-16; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Other Acute Postoperative Pain
Keywords: Pediatric spinal anesthesia, paracetamol, dipyrone
MeSH Terms: interventions — Acetaminophen; Dipyrone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Active Comparator): 15 mg/kg paracetamol, IV (in the vein)(premixed with 0.9% sodium chloride to a total of 50 ml)single dose
  Interventions: Drug: Paracetamol
- Dipyrone (Active Comparator): 15 mg/kg IV (in the vein)dipyrone received (premixed with 0.9% sodium chloride to a total of 50 ml), single dose
  Interventions: Drug: Dipyrone

INTERVENTIONS:
Drug: Paracetamol — 15 mg/kg IV (premixed with 0.9% sodium chloride to a total of 50 ml), preoperative single dose
  Other Names: Parol
  Arms: Paracetamol
Drug: Dipyrone — 15 mg/kg IV (premixed with 0.9% sodium chloride to a total of 50 ml), preoperative single dose
  Other Names: Metamizole
  Arms: Dipyrone

SUMMARY:
We conducted a prospective, randomized double-blind study to compare the effectiveness of intravenous paracetamol and dipyrone for preventing pain during early postoperative period in school-age children undergoing lower abdominal surgery with spinal anesthesia.

DETAILED DESCRIPTION:
The intensity of postoperative pain was assessed using a visual analog scale (VAS) (0 represented no pain and 10 the worst pain ever experienced) at 15, 30, 60th minutes, and 2nd, 4th, 6th hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status I and II children undergoing elective lower abdominal surgery

Exclusion Criteria:

* increased intracranial pressure hemorrhagic diathesis infection at the puncture site Those with a known history of allergy to the study drugs

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from pain intensity until postoperative 6 hours | Pain intensity recorded until postoperative 6 hours
  The intensity of postoperative pain was assessed using a visual analog scale (VAS) (0 represented no pain and 10 the worst pain ever experienced) at 15, 30, 60th minutes, and 2nd, 4th, 6th hours postoperatively.

REFERENCES:
- [Derived] Caliskan E, Sener M, Kocum A, Ozyilkan NB, Ezer SS, Aribogan A. The efficacy of intravenous paracetamol versus dipyrone for postoperative analgesia after day-case lower abdominal surgery in children with spinal anesthesia: a prospective randomized double-blind placebo-controlled study. BMC Anesthesiol. 2013 Oct 22;13(1):34. doi: 10.1186/1471-2253-13-34. PMID 24144215